CLINICAL TRIAL: NCT06912529
Title: Axicabtagene Ciloleucel CAR T-cells in Patients With Relapsed or Refractory Primary Mediastinal B-cell Lymphoma
Acronym: PRIME-CAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder of the study terminated contract
Sponsor: Universität Münster (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniMS23_0018; 2024-510972-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: B-cell Lymphoma Refractory; B-cell Lymphoma Recurrent
MeSH Terms: interventions — Leukapheresis; Blood Component Removal; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): While completing the screening process corticoid therapy may be continued up 7 days prior to leukapheresis. After leukapheresis, one cycle of any therapy can be given as bridging therapy to reduce tumor burden if clinically necessary. Lymphodepletion (LD) can be started after PET-CT-based staging. LD consists of lymphocyte depleting chemotherapy with fludarabine and cyclophosphamide (FC) applied on day -5 to day -3 followed by administration of axicabtagene ciloleucel on day 0. Patients will be observed as inpatients until at least day 10. Once the patient is discharged, outpatient visits including PET-CT-based staging are required on day 30 (±2 days), day 100 (±7 days), month 6 and 12 after axicabtagene ciloleucel administration.
  Interventions: Procedure: Leukapheresis; Drug: Bridging Therapy; Drug: Lymphodepletion; Genetic: Axicabtagene Ciloleucel

INTERVENTIONS:
Procedure: Leukapheresis — Axicabtagene ciloleucel is prepared from the patient's peripheral blood mononuclear cells, which are obtained via a standard leukapheresis procedure.
  Other Names: apheresis
Drug: Bridging Therapy — Bridging therapy refers to treatment used to control a patient's disease or disease related inflammation prior to lymphodepletion.
Drug: Lymphodepletion — Patients will receive a non-myeloablative lymphodepleting regimen consisting of fludarabine and cyclophosphamide (FC) to induce lymphocyte depletion and create an optimal environment for expansion of axicabtagene ciloleucel in vivo.
Genetic: Axicabtagene Ciloleucel — Patient will receive the axicabtagene ciloleucel infusion in the hospital followed by daily monitoring in the hospital.
  Other Names: axi-cel

SUMMARY:
This phase II study will evaluate the efficacy, safety and tolerability of second-line treatment with axicabtagene ciloleucel in primary mediastinal B-cell lymphoma patients (PMBCL).

DETAILED DESCRIPTION:
Patients who are refractory or relapse after first-line therapy of PMBCL have poor outcomes when treated with standard salvage therapy consisting of high-dose therapy and autologous stem cell transplantation. Recent studies and real-world data on CAR T-cells in patients with early relapsed or refractory aggressive B-cell lymphoma, particularly diffuse large cell B-Cell lymphoma, showed improved event free survival and overall survival with axicabtagene ciloleucel compared with the previous standard of care. These reports suggest comparable efficacy with similar toxicity profiles for CAR T-cells in PMBCL. However, larger studies with CAR T-cells in patients who are refractory to first-line therapy or who relapse after an initial response are urgently needed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form (ICF) according to ICH/EU GCP and national regulations
2. Age > 18 years
3. ECOG performance status < 2
4. Histologically confirmed primary mediastinal B-cell lymphoma (PMBCL)

   * based on the 2022 World Health Organization (WHO) (R. Allagio et al.)
   * classification by local pathology laboratory assessment
5. Patients must have received adequate first-line therapy including:

   * An anti-CD20 monoclonal antibody (rituximab), and
   * CHOP or CHOP-like chemotherapy Note: CHOP-like chemotherapy corresponds to CHOEP, ACVBP or EPOCH or COPADEM. Patients who received dose-reduced CHOP (e.g., mini-CHOP) are excluded except for dose reductions of vincristine due to peripheral neuropathy. Patients who have received additional drugs in combination with CHOP or CHOP-like regimen are eligible.
6. Relapsed or refractory disease after first-line chemoimmunotherapy, documented by PET-CT:

   * Relapsed disease defined as complete remission to first-line therapy followed by biopsy-proven relapse
   * Refractory disease defined as:

     * Progressive disease (PD) during first-line therapy
     * Stable disease (SD) as best response after at least 4 cycles of first-line therapy (e.g., 4 cycles of R-CHOP) and biopsy-proven residual disease, or
     * Partial response (PR) as best response after at least 6 cycles, and biopsy-proven residual disease
7. At least 2 weeks must have elapsed since any prior systemic cancer therapy at the time the patient provides consent
8. Lymphoma tissue at recurrence available for central pathologic examination, exploratory endpoints, and ancillary studies (detailed sample collection requirements are described in protocol section 8.2)
9. Patients must have at least 1 measurable lesion per the Lugano Classification on anatomical imaging such as computed tomography (CT) imaging (functional imaging such as PET may not be used to identify a measurable lesion). A measurable lesion is defined as greater than 1.5 cm LDi for lymph node and greater than 1.0 cm LDi for extranodal lesions
10. Patients must be eligible for CAR T-cells as defined by:

    * Patient deemed eligible for CAR T-cells therapy by the study physician
    * Adequate vascular access for leukapheresis procedure (either peripheral or central venous line)
11. Adequate bone marrow, renal, hepatic, cardiac and pulmonary function defined as:

    * Absolute neutrophil count (ANC) ≥ 1000 cells/μL
    * Absolute lymphocyte count > 100/μL
    * Platelets ≥ 75,000 cells/μL
    * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 40 ml/min
    * Transaminases (AST and ALT) <2.5 x ULN
    * Total bilirubin < 1.5 x ULN unless other reason known (Gilbert-Meulengracht-Syndrome in which 3 x ULN would be acceptable)
    * Left ventricular ejection fraction (LVEF) ≥ 40% and no evidence of clinically significant pericardial effusion, and no significant abnormal electrocardiogram (ECG) findings
    * No evidence of Grade 2 (per Common Terminology Criteria for Adverse Events [CTCAE] 5.0) or greater pleural effusion or ascites (subjects with Grade 1 ascites or pleural effusion are eligible)
    * Baseline oxygen saturation > 92% on room air
12. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 12 months are not considered to be of childbearing potential)
13. Sexually active men and FCBP must agree to use one of the highly effective contraceptive methods (combined oral contraceptives using two hormones, contraceptive implants, injectables, intrauterine devices, sterilized partner) together with one of the barrier methods (latex condoms, diaphragms, contraceptive caps) while on study; this should be maintained for 12 months after the last dose of study drug
14. Willingness not to drive a vehicle for 8 weeks post CAR T-cell treatment

Exclusion Criteria:

1. Patients who received more than one prior line of systemic therapy
2. Prior CD19-targeted therapy
3. History of another primary malignancy that has not been in remission for at least 2 years (except for non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast)). A maintenance treatment is not allowed
4. History or presence of non-malignant CNS disorder, such as seizure disorder requiring anti-convulsive therapy, cerebellar disease, any autoimmune disease with CNS involvement, posterior reversible encephalopathy syndrome (PRES), or cerebral edema with confirmed structural defects by appropriate imaging. History of stroke or transient ischemic attack within 12 months prior to enrollment.

   • Secondary CNS involvement of PMBCL is not an exclusion criterion
5. History of acute or chronic active hepatitis B or C infection. If there is a positive history of treated hepatitis B or hepatitis C, the viral load must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing
6. Positive for human immunodeficiency virus (HIV) unless taking appropriate anti-HIV medications, with an undetectable viral load by PCR and with a CD4 count > 200 cells/μl
7. Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal catheter). Dedicated venous access catheters, such as a Port-a-Cath or Hickman catheter, are permitted
8. Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antimicrobials at the time of enrollment
9. Presence of cardiac atrial or ventricular lymphoma involvement
10. History of any one of the following cardiovascular conditions within the past 12 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
11. History of any medical condition including but not limited to autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression and/or systemic disease modifying agents within the last year. Endocrine conditions that require maintenance with physiologic dose steroids are allowed
12. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed
13. History of severe immediate hypersensitivity reaction to any of the agents used in this study, including aminoglycosides, cyclophosphamide, fludarabine or tocilizumab
14. Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study
15. FCBP who are pregnant or breastfeeding
16. In the investigator's judgment, the patient is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
17. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness.
18. Simultaneously active participation in another clinical trial involving an IMP within 30 days prior to enrolment into this clinical trial
19. Patients with a physical or psychiatric condition which at the investigator's discretion may put the patient at risk, may confound the trial results, or may interfere with the patient's participation in this clinical trial
20. Known or persistent abuse of medication, drugs or alcohol
21. History of deep vein thrombosis or pulmonary embolism requiring therapeutic anticoagulation within 6 months of enrollment
22. Primary immunodeficiency
23. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
24. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Complete metabolic response (CMR) | 3 months from axicabtagene ciloleucel infusion
  Complete metabolic response at 3 months from axicabtagene ciloleucel infusion (without additional anticancer therapy). Assessment of response will be based on the Lugano classification.

SECONDARY OUTCOMES:
Best response rate | between day 30 and 12 months from axicabtagene ciloleucel infusion
  Best response rate is defined as the percentage of responder determined investigator disease assessment (INV) among all patients between day 30 and 12 months from axicabtagene ciloleucel infusion.
Duration of complete metabolic response (DOCMR) | 3 months from axicabtagene ciloleucel infusion
  The time from attainment of CMR to the date of first documented disease progression/relapsed (based on investigator disease assessment (INV)) or lymphoma-related deaths
Time to first response | time from axicabtagene ciloleucel infusion after which the first response (CMR without additional anticancer therapy/PMR at 30 days, 3 months, 6 months and 12 months) has ocurredhas occurred
  Time from axicabtagene ciloleucel infusion after which the first response (CMR without additional anticancer therapy/PMR at day 30, 3 months, 6 months, 12 months) has ocurred
Relapse rate (RR) | 3 months from axicabtagene ciloleucel infusion
  Number of relapses divided by the number of patients included with complete metabolic response (CMR) at 3 months from axicabtagene ciloleucel infusion (without additional anticancer therapy) based on investigator disease asessment (INV)
Progression-free survival (PFS) | until last visit of patient, assessed up to 24 months
  Time from enrolment to the first observation of documented disease progression/relapsed (based on INV) or death due to any cause
Progression-free survival modified (mPFS) | until last visit of patient, assessed up to 24 months
  Time from axicabtagene ciloleucel infusion to the first observation of documented disease progression/relapsed (based on INV)) or death due to any cause
Event-free survival (EFS) | until last visit of patient, assessed up to 24 months
  Time from enrolment to failure to achieve a CMR at 12 months post CAR infusion, or start of any new lymphoma therapy, or the first observation of documented disease progression/relapsed (based on INV)) or death due to any cause, whichever comes first.
Modified EFS (mEFS) | until last visit of patient, assessed up to 24 months
  Time from axicabtagene ciloleucel infusion to failure to achieve a CMR at 12 months post CAR infusion, or start of any new lymphoma therapy, or to the first observation of documented disease progression/relapsed (based on INV)), or death due to any cause, whichever comes first.
Overall survival (OS) | From enrollment to the date of death. Alive patients will be censored at the last date where it is known that the patient is still alive, assessed up to 24 months
  Time from enrolment to the date of death from any cause.
Overall survival modified (mOS) | From date of axicabtagene ciloleucel infusion to the date of death. Alive patients will be censored at the last date where it is known that the patient is still alive, assessed up to 24 months
  From date of the axicabtagene ciloleucel infusion to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lenz, Prof, Study Director — Universität Münster
Locations (1):
- Medizinische Klinik A Hämatologie, Hämostaseologie, Onkologie und Pneumologie Universitätsklinikum Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No